CLINICAL TRIAL: NCT03215160
Title: Effectiveness of Mobilization Exercises on Total Knee Arthroplasty Rehabilitation
Brief Title: Using Mobilization Exercises on Total Knee Arthroplasty Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Sezen Karabörklü Argut, MSc Research Assistant, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22595
Record Dates: First submitted 2017-06-19; First posted 2017-07-12 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Total Knee Arthroplasty; Total Knee Replacement
Keywords: Mobilization; Manual Therapies; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobilization Exercise Group (Experimental): Mobilization exercises in addition to classical exercises performed in the early post-op period
  Interventions: Behavioral: Exercises
- Classical Exercise Group (Active Comparator): only classical exercises performed in the early post-op period
  Interventions: Behavioral: Exercises

INTERVENTIONS:
Behavioral: Exercises — mobilization exercises (Patellofemoral joint, Tibiofemoral joint, Soft tissue) and classical exercises performed in the early post-op period

SUMMARY:
There is no definite evidence about the most effective treatment approach in early-stage rehabilitation after total knee arthroplasty surgery. The purpose of this study is to investigate the effects of mobilization exercises applied with classical exercises on pain, joint range of motion, edema, function, quality of life and patient satisfaction in early stage rehabilitation after total knee arthroplasty surgery.

DETAILED DESCRIPTION:
There is no definite evidence about the most effective treatment approach in early-stage rehabilitation after total knee arthroplasty surgery. The purpose of this study is to investigate the effects of mobilization exercises applied with classical exercises on pain, joint range of motion, edema, function, quality of life and patient satisfaction in early stage rehabilitation after total knee arthroplasty surgery. Patients with bicompartmental total knee arthroplasty operation due to knee osteoarthritis will randomly assign to 2 groups. Patients in group 1 will treat with mobilization exercises in addition to classical exercises performed in the early post-op period; patients in group 2 will treat only with classical exercises.

ELIGIBILITY:
Inclusion Criteria:

* Patients with TKA surgery due to the diagnosis of knee OA
* Between the ages of 50-75 years

Exclusion Criteria:

* Revision TKA,
* Previous unicompartmental arthroplasty or tibial osteotomy,
* Hemophilia,
* Rheumatic diseases,
* Lower extremity fractures and tumors,
* Neurological diseases leading to muscle weakness in the lower limbs,
* Patients with emotional and cognitive problems

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-07-22 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Range of Motion Degree at 2 weeks | Baseline, Post-op 2 weeks, and Post-op 2 months
  Passive knee flexion range of motion

SECONDARY OUTCOMES:
Change from Baseline Pain Degree at 2 weeks | Baseline, Post-op 2 weeks, and Post-op 2 months
  Patient reported pain degree
Function | Baseline, Post-op 2 weeks, and Post-op 2 months
  Functional Performance tests

OTHER OUTCOMES:
Satisfaction levels of the patients | At 2 months
  Satisfaction levels of the patients with Global Rating of Change Score

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Harvey LA, Brosseau L, Herbert RD. Continuous passive motion following total knee arthroplasty in people with arthritis. Cochrane Database Syst Rev. 2014 Feb 6;2014(2):CD004260. doi: 10.1002/14651858.CD004260.pub3. PMID 24500904
- [Background] Cross M, Smith E, Hoy D, Nolte S, Ackerman I, Fransen M, Bridgett L, Williams S, Guillemin F, Hill CL, Laslett LL, Jones G, Cicuttini F, Osborne R, Vos T, Buchbinder R, Woolf A, March L. The global burden of hip and knee osteoarthritis: estimates from the global burden of disease 2010 study. Ann Rheum Dis. 2014 Jul;73(7):1323-30. doi: 10.1136/annrheumdis-2013-204763. Epub 2014 Feb 19. PMID 24553908
- [Background] Nelson AE, Allen KD, Golightly YM, Goode AP, Jordan JM. A systematic review of recommendations and guidelines for the management of osteoarthritis: The chronic osteoarthritis management initiative of the U.S. bone and joint initiative. Semin Arthritis Rheum. 2014 Jun;43(6):701-12. doi: 10.1016/j.semarthrit.2013.11.012. Epub 2013 Dec 4. PMID 24387819
- [Background] Jacobs CA, Christensen CP. Factors influencing patient satisfaction two to five years after primary total knee arthroplasty. J Arthroplasty. 2014 Jun;29(6):1189-91. doi: 10.1016/j.arth.2014.01.008. Epub 2014 Jan 21. PMID 24534535
- [Background] Bade MJ, Kohrt WM, Stevens-Lapsley JE. Outcomes before and after total knee arthroplasty compared to healthy adults. J Orthop Sports Phys Ther. 2010 Sep;40(9):559-67. doi: 10.2519/jospt.2010.3317. PMID 20710093
- [Background] Noble PC, Gordon MJ, Weiss JM, Reddix RN, Conditt MA, Mathis KB. Does total knee replacement restore normal knee function? Clin Orthop Relat Res. 2005 Feb;(431):157-65. doi: 10.1097/01.blo.0000150130.03519.fb. PMID 15685070
- [Background] Ebert JR, Munsie C, Joss B. Guidelines for the early restoration of active knee flexion after total knee arthroplasty: implications for rehabilitation and early intervention. Arch Phys Med Rehabil. 2014 Jun;95(6):1135-40. doi: 10.1016/j.apmr.2014.02.015. Epub 2014 Mar 3. PMID 24602550
- [Background] Bade MJ, Stevens-Lapsley JE. Early high-intensity rehabilitation following total knee arthroplasty improves outcomes. J Orthop Sports Phys Ther. 2011 Dec;41(12):932-41. doi: 10.2519/jospt.2011.3734. Epub 2011 Sep 30. PMID 21979411
- [Derived] Karaborklu Argut S, Celik D, Kilicoglu OI. The Combination of Exercise and Manual Therapy Versus Exercise Alone in Total Knee Arthroplasty Rehabilitation: A Randomized Controlled Clinical Trial. PM R. 2021 Oct;13(10):1069-1078. doi: 10.1002/pmrj.12542. Epub 2021 Feb 3. PMID 33352007